CLINICAL TRIAL: NCT01299649
Title: A Retrospective Observational Database Study To Compare In-Hospital All-Cause Mortality in Critically Ill Patients Undergoing Echocardiography With or Without DEFINITY®
Brief Title: Retrospective Safety Study to Compare Mortality in Intensive Care Unite (ICU) Patients Undergoing Echocardiography With or Without DEFINITY®
Acronym: DEF-418
Status: Completed | Type: Observational
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Other Study IDs: DMP 115-418
Record Dates: First submitted 2011-02-16; First posted 2011-02-18 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2011-02

CONDITIONS: Cardiovascular Disease
Keywords: CAD
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-contrast echocardiography: Non-contrast echocardiography
- Contrast Echocardiography: Contrast Echocardiography

SUMMARY:
Retrospective analysis to observe changes in short term mortality

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* At least 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All that received an echocardiogram
Sampling Method: Non-Probability Sample
Enrollment: 4300000 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Short term mortality | 48 hours post echo produre

CONTACTS AND LOCATIONS:
Locations (1):
- Lantheus Medical Imaging, North Billerica, Massachusetts, United States